CLINICAL TRIAL: NCT03362424
Title: Mesenchymal Stem Cells in Rotator Cuff Repair - a Randomized Prospective Study
Brief Title: Mesenchymal Stem Cells in Rotator Cuff Repair
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Cryogenesis company stopped supplying mesenchymal cells
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Eduardo Angeli Malavolta, Principal investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2.335.243
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Rotator Cuff Tear; Tendon Injuries; Mesenchymal Stem Cell
MeSH Terms: conditions — Rotator Cuff Injuries; Tendon Injuries

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Surgeon and patients not blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenchymal stem cell group (Experimental): rotator cuff repair stem cells
  Interventions: Biological: Mesenchymal stem cell; Procedure: Rotator cuff repair
- Control group (Active Comparator): rotator cuff repair
  Interventions: Procedure: Rotator cuff repair

INTERVENTIONS:
Biological: Mesenchymal stem cell — Mesenchymal stem cells applies at the end of rotator cuff repair in de active group
  Arms: Mesenchymal stem cell group
Procedure: Rotator cuff repair — Rotator cuff repair

SUMMARY:
Randomized clinical study involving 44 patients, evaluating the effect of mesenchymal cells on rotator cuff repair. The primary outcome will be post-operative MRI tendon integrity and secondary outcomes clinical assessment by the UCLA and American Shoulder and Elbow Surgeons (ASES) scales and pain by visual analog scale (VAS).

DETAILED DESCRIPTION:
Rotator cuff tendinopathy is the main cause of shoulder pain and tear of these tendons affects 20% of the population. Although arthroscopic repair leads to satisfactory clinical results, the retear rates varies from 4 to 94%. The main cause of failure after rotator cuff repair is not related to the material used, but to the tissue deficiency and the healing process between the tendon and the bone. After the intervention, the rotator cuff does not restore its original histological characteristics and its fixation occurs through scar tissue with lower biomechanical resistance. There are few clinical studies on the use of mesenchymal cells in rotator cuff repair,, with good results.

The investigators will perform a randomized clinical study involving 44 patients, evaluating the effect of mesenchymal cells on rotator cuff repair. The primary outcome will be post-operative MRI tendon integrity and secondary outcomes clinical assessment by the UCLA and American Shoulder and Elbow Surgeons (ASES) scales and pain by visual analog scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Full thickness posterosuperior rotator cuff tear, of small or medium size, fully repairable at the time of surgery, regardless of size;
* Pain and / or decreased shoulder function for at least 3 months, with no improvement with non-surgical treatment;
* Absence of the following changes in MRI:
* Fat degeneration of the rotator cuff musculature of grade 3 according to the classification of Fuchs (presence of equal or superior amount of fat compared to muscle fibers);
* Absence of the following changes in radiographs
* Advanced glenohumeral arthrosis (grades 2, 3 and 4 of Samilson and Prieto
* Signs of rotator cuff arthropathy, according to Seebauer classification;
* Skeletal maturity;
* Absence of surgeries or previous fractures in the shoulder in question;
* Absence of psychiatric illnesses, fibromyalgia or painful pathologies of the cervical spine;
* Absence of rheumatic diseases or chronic use of corticosteroids;
* Absence of active or recent infection;
* Absence of thrombocytopenia, coagulopathies or chronic use of anticoagulants;
* Absence of vascular or neurological lesions affecting the upper limb;
* Absence of pregnancy;
* Clinical non-compensated comorbidities;
* Chronic use of corticosteroids;
* Consent to free and informed consent;
* Live in Brazil.

Exclusion Criteria:

* Visualization during the operative event of one or more of the findings:
* Irreparable rupture of rotator cuff;
* Subsecapularis tear involving two thirds or more of its extension;
* Need to open surgery.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
MRI integrity | 6 months
  Sugaya classification

SECONDARY OUTCOMES:
American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASES) | 6, 12 and 24-months
  minimum 0 points, maximum 100 points. Higher values are considered best outcomes.
University at California at Los Angeles Shouder Rating Scale (UCLA) | 6, 12 and 24-months
  minimum 3 points, maximum 35 points. Higher values are considered best outcomes.
Visual Analog Scale for Pain (VAS) | 6, 12 and 24-months
  miminum 0 points, maximum 10 points. Higher values are considered worst outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: EDUARDO ANGELI MALAVOLTA A Malavolta, PhD, Principal Investigator — MD, PhD, Associate Professor
Locations (1):
- Universidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided